CLINICAL TRIAL: NCT06296290
Title: Impact of Prolonged Cold-water Swimming on Heart Rate and Cardiac Function in Healthy Swimmers.
Brief Title: Impact of Prolonged Cold-water Swimming on Heart Rate and Cardiac Function
Acronym: CARDIOCOLD
Status: Completed | Type: Observational
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: CARDIOCOLD
Record Dates: First submitted 2024-02-29; First posted 2024-03-06 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-02

CONDITIONS: Hypothermia
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All participants: The participants are the swimmers engaged in the 6-hour cold water swim during the Channel Swim Camp who volunteered to participate in the study.

SUMMARY:
A significant medical risk associated with hypothermia during exercise in a cold environment cardiac arrhythmia due to a possible autonomic conflict. However, little is known about the changes in heart rate and cardiac function after prolonged cold water swimming.

The investigators propose to measure the changes in core temperarure during and after a cold water swim at at a water temperature below 15.5°C qualifying for English Channel swim and to test the association with changes in heart rate variability, resting electrocardiogram and left ventricle function.

ELIGIBILITY:
Inclusion Criteria:

* swimmers taking part in the Channel Swim Camp
* swimmers above 18 years of age
* swimmers willing and able to give informed consent for participation in the study

Exclusion Criteria:

* swallowing disorder
* chronic gastrointestinal disease
* MRI scheduled within 48 hours after the race.
* known cardiac arythmia or cardiovascular disease

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Swimmers participating in the 6-hour cold-water swim, qualifying for the English Channel swim at the Channel Swim Camp (Dinard, France).
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2022-06-04 (Actual); Primary Completion 2022-06-06 (Actual); Study Completion 2022-08-15 (Actual)

PRIMARY OUTCOMES:
Heart rate from a resting ECG recording | Two Time points (1) the day before the race and (2) at 30 min after ending the race
  Waves, intervals & segments of the normal ECG trace was collected
Heart rate from a 5-minute ECG recording | Two Time points (1) the day before the race and (2) at 30 min after ending the race
  Heart rate variability (HRV) parameters including time-domain measures and frequency-time measures
Transthoracic echocardiography (TTE) analysis | Two Time points (1) the day before the race and (2) at 30 min after ending the race
  Left and right ventricular and atrial dimensions, and systolic and diastolic ventricular function assessment were collected
Change in Body Core Temperature | Time Frame: Continuous measurement was collected from 30 minutes before the race until 2 hours after the end of the race for each swimmer]
  Measurement of Body Core Temperature using an ingestible electronic sensor (e-Celsius®, BodyCap , Caen, France) which provide a continuous validated measurement

SECONDARY OUTCOMES:
Body composition, body fat mass | One measurement assessed the day before the race
  Fat mass (in kg, % of body mass [fat mass and body mass were combined to report % of body mass) was measured using bioelectrical impedance analysis (mBCA 525, Seca, Germany).
Body composition, fat-free mass | One measurement assessed the day before the race
  Fat-free mass (in kg, % of body mass [fat-free mass and body mass were combined to report % of body mass) was measured using bioelectrical impedance analysis (mBCA 525, Seca, Germany).
Duration | The duration of swimming was collected from the organisers immediately after the race
  Duration of the swimming
Individual characteristics, gender | One evaluation assessed the day before the race
  The variable collected was the gender of participants
Individual characteristics, age | One evaluation assessed the day before the race
  The variable collected was the age of participants
Individual characteristics, training in cold environment | One evaluation assessed the day before the race
  The variable collected was the type of specific training in cold environment (yes/no)

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Caen Normandie, Caen, France

IPD SHARING:
Plan to Share IPD: Undecided